CLINICAL TRIAL: NCT06727214
Title: Survival Benefit of Neoadjuvant Systemic Chemotherapy in Muscle Invasive Bladder Cancer and Factors Affecting Its Response - Retrospective Study
Brief Title: Survival Benefits of Neoadjuvant Systemic Chemotherapy in Muscle Invasive Bladder Cancer
Acronym: AssiutU
Status: Not yet recruiting | Type: Observational
Sponsor: Sara Mahmoud Ahmed Mahmoud (Other)
Responsible Party: Sponsor-Investigator, Sara Mahmoud Ahmed Mahmoud, doctor, Assiut University
Organization: Assiut University (Other)
Other Study IDs: Survival of NAC in MIBC
Record Dates: First submitted 2024-12-03; First posted 2024-12-10 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2024-12

CONDITIONS: Bladder Urothelial Carcinoma
Keywords: survival benefits; neoadjuvant CTH; bladder cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Drug Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- MIBC patients who received NAT: muscle invasive bladder cancer patients who received neoadjuvant chemotherapy
  Interventions: Drug: Chemotherapy with platine

INTERVENTIONS:
Drug: Chemotherapy with platine — medical records that patients received neoadjuvant systemic chemotherapy platine based

SUMMARY:
Muscle-invasive bladder cancer (MIBC) is an aggressive disease with a high-risk of early metastasis and cancer specific mortality. The gold standard treatment of MIBC is radical cystectomy (RC) in conjunction with concomitant bilateral pelvic lymphadenectomy . While radical cystectomy remains a primary management strategy for MIBC, high rates of recurrence with surgery alone highlight the likelihood of occult micrometastatic disease at the time of diagnosis. Due to the development and implementation of neoadjuvant chemotherapy prior to radical cystectomy, the prognosis for MIBC patients undergoing radical cystectomy has improved .

DETAILED DESCRIPTION:
The goals of neoadjuvant chemotherapy administration are to; eradicate the micro-metastases, avoid the release and implantation of malignant cells during cystectomy, and extend the survival of these patients.

Clinical trial data supports the use of neoadjuvant platinum-based chemotherapy for patients with non-metastatic MIBC. Based on Level I evidence, use of preoperative platinum based chemotherapy is now included in the guideline recommendations from the American Urologic Association (AUA), American Society of Clinical Oncology (ASCO), National Comprehensive Cancer Network (NCCN), and European Association of Urology (EAU) . In the Southwest Oncology Group (SWOG) Intergroup study, RC alone was compared with three cycles of neoadjuvant MVAC (methotrexate, vinblastine, doxorubicin, and cisplatin), followed by radical cystectomy. This randomized trial showed that the median survival duration was 77 months in patients with combination treatment, and 46 months in patients with upfront RC alone.

ELIGIBILITY:
Inclusion Criteria:

* Age >18
* histological proven MIBC patient treated with neoadjuvant systemic chemotherapy( platinum based )

Exclusion Criteria:

* Non muscle invasive bladder cancer (NMIBC)
* Metastatic patients
* Patients treated with surgery firstly

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Data Record of the patients will be reviewed for the following : *Clinical features:Age , Sex , Smoking ,base line renal function , comorbidities *HistoPathological features: Histological type of bladder cancer ,Carcinoma in situ,Lymphovascular invasion ( LVI)
  * Type of neoadjuvant chemotherapy received: Platinum based ( cisplatin, carboplatin)
  * Number of cycles .
  * Response to neoadjuvant chemotherapy : Assesed by radiological tools ( MRI , CT ) according to Recist criteria.
  * Follow up after finishing the course of neoadjuvant chemotherapy , using imaging and examination to detect the response and survival outcomes.
Sampling Method: Probability Sample
Enrollment: 87 (Estimated)
Dates: Start 2025-11-04 (Estimated); Primary Completion 2026-11-04 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Evaluating the factors affecting the response of neoadjuvant chemotherapy in muscle invasive bladder cancer | 3 to 6 months (from previous medical reports )
  evaluating the neoadjuvant respose by clinical examination and radiological tools ( CT , MRI ) according to Recist criteria

SECONDARY OUTCOMES:
Disease free survival (DFS) | thorough study completion (an average 1 year )
  DFS the length of time after primary treatment for a cancer ends that the patient survives without any signs or symptoms of that cancer.
overall survival (OS) | from the randomization until the date of 1st decument progression or death from any cause , whichever come first assesed up to 100 weeks
  OS: defined as the length of time from either the date of diagnosis or the start of treatment for cancer, that patients are still alive.
Progression Free Survival ( PFS ) | an average 2 years
  the average lenght of time after the start of treatment in which a person is alive and their cancer does not grow or spread

CONTACTS AND LOCATIONS:
Overall Officials: Rehab Farouk Mohamed, Professor, Study Director — Assiut University

REFERENCES:
- [Background] Advanced Bladder Cancer (ABC) Meta-analysis Collaboration. Neoadjuvant chemotherapy in invasive bladder cancer: update of a systematic review and meta-analysis of individual patient data advanced bladder cancer (ABC) meta-analysis collaboration. Eur Urol. 2005 Aug;48(2):202-5; discussion 205-6. doi: 10.1016/j.eururo.2005.04.006. Epub 2005 Apr 21. PMID 15939524
- [Background] Motterle G, Andrews JR, Morlacco A, Karnes RJ. Predicting Response to Neoadjuvant Chemotherapy in Bladder Cancer. Eur Urol Focus. 2020 Jul 15;6(4):642-649. doi: 10.1016/j.euf.2019.10.016. Epub 2019 Nov 8. PMID 31708469
- [Background] Daneshmand S, Nazemi A. Neoadjuvant Chemotherapy in Variant Histology Bladder Cancer: Current Evidence. Eur Urol Focus. 2020 Jul 15;6(4):639-641. doi: 10.1016/j.euf.2020.04.011. Epub 2020 May 22. PMID 32451316
- [Background] Hu J, Chen J, Ou Z, Chen H, Liu Z, Chen M, Zhang R, Yu A, Cao R, Zhang E, Guo X, Peng B, Deng D, Cheng C, Liu J, Li H, Zou Y, Deng R, Qin G, Li W, Wang L, Chen T, Pei X, Gong G, Tang J, Othmane B, Cai Z, Zhang C, Liu Z, Zu X. Neoadjuvant immunotherapy, chemotherapy, and combination therapy in muscle-invasive bladder cancer: A multi-center real-world retrospective study. Cell Rep Med. 2022 Nov 15;3(11):100785. doi: 10.1016/j.xcrm.2022.100785. Epub 2022 Oct 19. PMID 36265483
- [Background] Yin M, Joshi M, Meijer RP, Glantz M, Holder S, Harvey HA, Kaag M, Fransen van de Putte EE, Horenblas S, Drabick JJ. Neoadjuvant Chemotherapy for Muscle-Invasive Bladder Cancer: A Systematic Review and Two-Step Meta-Analysis. Oncologist. 2016 Jun;21(6):708-15. doi: 10.1634/theoncologist.2015-0440. Epub 2016 Apr 6. PMID 27053504